CLINICAL TRIAL: NCT00932594
Title: Create the New Serial Treatment of Temporomandibular Disorders
Brief Title: The New Serial Treatment of Temporomandibular Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, zhang zhiguang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSU-5010
Record Dates: First submitted 2009-06-29; First posted 2009-07-03 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Temporomandibular Disorder
Keywords: Create the New Serial Treatment of TMD; Promote the Classification of Biodynamics in the TMD; Evaluate the Effect of Adjusting TMJ Treatment; Establish the New Standard of the TMJ Treatment; Invent New Device to Measure Pressure without Trauma
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 1.Arthrocentesis only (Active Comparator): Patients only have Arthrocentesis, but without adjusting the pressure of the TMJ
  Interventions: Other: Do not adjust the pressure of TMJ
- 3.Arthroscopic Treatment (Active Comparator): Patient receives Arthroscopic treatments without adjusting the TMJ pressure
  Interventions: Other: Do not adjust the pressure of TMJ
- 4.Arthroscopic with Adjust Pressure (Active Comparator): Arthroscopic Treatment with Adjust TMJ Pressure Treatment, during the Arthroscopic treatment adjust the pressure of TMJ to normal value
  Interventions: Procedure: Adjust the TMJ Pressure to Normal Value
- 5.The TMJ Orperation Treatment (Active Comparator): The TMJ Operation Treatment without adjusting the pressure of TMJ
  Interventions: Other: Do not adjust the pressure of TMJ
- 6.The TMJ Operation with Adjust Pressure (Active Comparator): The TMJ Operation with Adjust TMJ Pressure Treatment, during the treatments to adjust the TMJ pressure to normal value
  Interventions: Procedure: Adjust the TMJ Pressure to Normal Value
- 7.Bite Plate Treatment (Active Comparator): Bite Plate Treatment for Temporomandibular Disorders without adjusting the pressure of TMJ
  Interventions: Other: Do not adjust the pressure of TMJ
- 8.Bite Plate with Adjust pressure (Active Comparator): Bite Plate and Adjust Pressure Treatment for Temporomandibular Disorders, during the treatments adjust the pressure of TMJ to normal value
  Interventions: Procedure: Adjust the TMJ Pressure to Normal Value
- 2.Arthrocentesis with adjust pressure (Active Comparator): Arthrocentesis with adjust pressure according to the pressure of TMJ
  Interventions: Procedure: Adjust the TMJ Pressure to Normal Value

INTERVENTIONS:
Procedure: Adjust the TMJ Pressure to Normal Value — Adjust the TMJ Pressure by the Operation Only Once for Each Patient
  Arms: 2.Arthrocentesis with adjust pressure; 4.Arthroscopic with Adjust Pressure; 6.The TMJ Operation with Adjust Pressure; 8.Bite Plate with Adjust pressure
Other: Do not adjust the pressure of TMJ — Do the treatments normally without additional treatment
  Arms: 1.Arthrocentesis only; 3.Arthroscopic Treatment; 5.The TMJ Orperation Treatment; 7.Bite Plate Treatment

SUMMARY:
The purpose of this study is to look at temporomandibular joint (TMJ) pressure as a guideline to analyze the different treatments for temporomandibular disorder (TMD), and judge the feasibility of the adjust TMJ pressure treatment and to reach a conclusion on the different treatments for different types of TMD, and determine the new serial treatment of temporomandibular disorders.

DETAILED DESCRIPTION:
Temporomandibular Disorder is a common disease nowadays, but there is no guideline for the treatment of TMD. TMD can be divided into masticating muscles dysfunction; internal derangement; inflammation; osteoarthrosis, this study will classify the internal derangement, inflammation and osteoarthrosis into three types according to the TMJ pressure. Then the patient will receive the adjust pressure treatment according to their TMJ pressure. The first part of the TMD patients will receive psychogenic treatment, medicine, physical treatment, bite plate, occlusion treatment, rebuilding occlusion treatment, orthodontic treatment, et. If the patients do not have a good curative effect, part of them will change the treatment into arthrocentesis, arthroscopic treatment or operation treatment, the other part of patients, according to their TMJ pressure, receiving the associated adjust pressure treatment or adjust pressure treatment only. This study will call on the patients for three years and collect the clinical information, then doing the medical statistics.

ELIGIBILITY:
Inclusion Criteria:

* Limited Month Opening
* Abnormal of the Month Opening Type
* Paint During the Month Open or Close
* Condylar Position Paint
* Clicking of the Temporomandibular Joint
* Enlargement of the Upper Temporomandibular Joint Gap
* Dislocation of the Temporomandibular Disc
* Bone of the Temporomandibular Joint Changement
* Patient in the Age of 16-60
* Voluntary Patient

Exclusion Criteria:

* Dysimmunity Disease
* Dysfunction of Heart Liver and Kidney Disease
* Patient can not do the Guide Line
* Life-threatening Patient
* Serious Limited Mouth Opening
* Epilepsy
* Tetanus
* Pregnancy or Women in the Pregnancy Period
* Supportive Temporomandibular Disease

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Estimated)
Dates: Start 2006-01; Primary Completion 2018-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: zg zhang, Master, Study Chair — GUANGHUA SHOOL OF STOMATOLOGY and HOSPITAL OF STOMATOLOGY SUN YAT-SEN UNIVERSITY
Locations (1):
- Guanghua School of Stomatology and Hospital of Stomatology, Guangzhou, Guangdong, China

REFERENCES:
- See also: The Web Site of the Guanghua College of Stomatology Sun Yat-sun University — http://www.zdkqyy.com